CLINICAL TRIAL: NCT02762734
Title: Multicenter Randomized Prevention Trial of Recurrence of Suicide Attempt by Adolescent by Sending SMS (MEDIACONNEX)
Brief Title: Prevention of Recurrence of Suicide Attempt by Adolescent by Sending SMS (MEDIACONNEX)
Acronym: MEDIACONNEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-A00744-45
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Suicide
Keywords: adolescent; suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDIA (Experimental): The patient will benefit of the usual care with additional text message (SMS or mail or other new media). The intervention for the group MEDIA is a "keeping in touch" intervention through sending of SMS (or mail or other new media). The patient will receive 6 SMS (or mail or other new media) during 6 months after the suicide attempt.
  Interventions: Other: MEDIA
- CLASSIC (No Intervention): The patient will benefit of the usual care.

INTERVENTIONS:
Other: MEDIA — The intervention for the group MEDIA is a "keeping in touch" intervention through sending of SMS (or mail or other new media). The patient will receive 6 SMS (or mail or other new media) during 6 months after the suicide attempt. The first one 7 days after the suicide attempt and the last one after 6 months. The first SMS (or mail or other new media) is sent soon after the suicide attempt because studies on adult suicide attempters underline the importance of an early start for the connectedness measures. The text message are evolving in time, and are adapted to the genre of the adolescent.
  Arms: MEDIA

SUMMARY:
MEDIACONNEX study propose a new way of connectedness for adolescents after a suicide attempt: it is based on the sending of SMS (or mail or other new media), over a period of 6 months after their suicide attempt (SA), in order to allow them to recourse to the care more easily and so to limit the risk of suicidal recurrence. The MEDIACONNEX study will be a multicenter controlled randomized trial (East of France) and there is a funding from the Hospital. The proposal trial will test the hypothesis that adolescent suicide attempters who are receiving SMS (or mail or other new media) from the unit of care in addition to the usual care will do less SA recurrence, than those who are receiving the usual care.

The primary objective is to determine whether the use of SMS (or mail or other new media) to keep in touch with adolescent suicide attempters in addition to the usual care, compare to usual care, will reduce the delay of recurrence of suicide attempt during 6 months after the SA.

DETAILED DESCRIPTION:
In industrialised countries, the incidence of SA among adolescents (ages 10-19 years old; 1) is estimated between 7% and 9% (2-3). Thirty percent of adolescents who have made a SA will do it again in the year. It appears that previous SA is "an independent and powerful predictor of futur attempt" (4). Moreover, one of the risk factors to commit suicide is to have made a SA, in particular during year preceding the suicide. To prevent suicide, it is thus important to prevent SA and particularly their recurrence. Research on adolescent suicide attempters focus in general on risk or protective factors (5-7). But despite of the knowledge on these characteristics, the rate of SA recurrence doesn't decrease. So, we have to be creative in the care proposals to limit it. An earlier study concluded that when adolescent suicide attempters were not any more in contact with the care system, they had more risk for SA recurrence (8). These last decades, news ways of care to prevent SA recurrence are developing for adults' suicide attempters on. These news cares may be divided into 2 categories: the "intensive cares" and the "connectedness" care (9). The intensive cares are for example specific therapies as cognitive-behaviour-therapy or dialectical behavior therapy (10-12), partial hospitalizations (13), brief psychological intervention at patients 'home (14)... And with some of these treatments, the rate or recurrence decreased (11-13). The "connectedness cares" are based on the fact of "keeping in touch" with patients and encouraging them to call in case of crises in order to avoid the recurrence. Motto and al. were the pioneer in the field of the connectedness in the 70s through the sending of letters regularly after the suicide attempt (15). It might be also through the sending of postcards (16-17), phone calls (18-19) or SMS (20)… As the intensive cares, these cares may have positive results on the rate of recurrence or on the numbers of recurrences. By the way, these different cares have diverse results depending sex or personality of patients (21). There is so a clinical relevance with the both sorts of cares but the "connectedness" one is easier to use, have a low cost and moreover, seems more appropriate for adolescents. Indeed, the therapeutic alliance with the young patients is not easy to install and an "intensive care" might be prevent them joining the care. Moreover, in another study in Nancy, France, the fact of being lost to follow-up by the caregivers is appeared as a risk factor of recurrence, even in 10-year after the suicide attempt. So, the fact of "keeping in touch" with adolescents after a suicide attempt is very important and they probably could accept easily this idea through one media they often use: short message system (SMS). There are yet some MobilHealth programs for adolescents as for adults in other specialties with good results (22-24).

MEDIACONNEX study also propose to assess the effectiveness of a new way of connectedness for adolescents after a SA : it is based on the sending of SMS (or mail or other new media), over a period of 6 months after their suicide attempt, in order to allow them to recourse to the care more easily and so to limit the risk of suicidal recurrence.

Design The MEDIACONNEX study is a simple blind, parallel group multisite randomized controlled trial which compares a program based on SMS (or mail or other new media) in addition to usual care (group MEDIA) to "only usual care" (group CLASSIC) provided to adolescents who attempted suicide and who were treated in-child and adolescent psychiatry unit at hospitals in the East of France. The comparison is based on rate of the recurrence suicide attempt between the two groups.

The primary objective is to determine whether the use of SMS (or mail or other new media) to keep in touch with adolescent suicide attempters in addition to the usual care, compare to usual care, will reduce the delay of recurrence of suicide attempt during 6 months after the SA.

Secondary objectives:

Determine whether the use of SMS (or mail or other new media) to keep in touch with adolescent suicide attempters in addition to the usual care, compare to usual care, will improve the evolution of their social network during 6 months Determine whether the use of SMS (or mail or other new media) to keep in touch with adolescent suicide attempters in addition to the usual care, compare to usual care, will improve the evolution of depression during 6 months Determine whether the use of SMS (or mail or other new media) to keep in touch with adolescent suicide attempters in addition to the usual care, compare to usual care, will improve the evolution of health-related quality of life during 6 months Determine the delay of recurrence of suicide attempt during 6 months after the end of the intervention by sending SMS (or mail or other new media) to evaluate if the intervention has an effect on the recurrence after stopped Determine the delay of death by suicide during 6 months after the end of the intervention by sending SMS (or mail or other new media) to evaluate if the intervention has an effect on the suicide after stopped Compare number of callphone spent in the unit of care between adolescents of the group Media and those of the group Classic

Participants Adolescent treated after a suicide attempt in a pediatric or psychiatric unit of the participating hospitals: Besançon, Dijon, Metz-Thionville, Nancy, Reims, and Strasbourg, FRANCE. The SA is defined as "a non-fatal act in which the individual liberally causes self-injury or ingests a substance in excess of any prescribed or generally recognised therapeutic dosage" (25). All the patients have a medical examination before the beginning of the research. Adolescent will be recruited during a psychiatric evaluation within 24 hours of admission to pediatric unit of the participating hospitals.

Inclusion Criteria:

To be 13-17 years old To be treated for a suicide attempt To have written consent of patient and his/her parents to participation in research

Non-inclusion Criteria:

The parents or/and patient who will refuse or who won't be able to accept to participate (somatic or understandability reasons), Incarcerated patient Those without any cell phone or any internet connexion or other new media.

Randomization The Zelen randomization will be used for this study (26-28). In each participating hospital, a member of the research team will screen each adolescent suicide attempters and when the adolescent suicide attempter will meet the eligibility criteria, his/her group for the study will be defined by a randomization. This patient will benefit of the usual care with additional SMS (group MEDIA) or of the usual care (group CLASSIC). Then, this member of the research will inform the adolescent 'psychiatrist who will present to the patient and his/her parents the design of the study, only for the group of the patient. The psychiatrist will also give information about the study and will gather an "informed consent".

Intervention The intervention for the group MEDIA is a "keeping in touch" intervention through sending of SMS (or mail or other new media). The patient will receive 6 SMS (or mail or other new media) during 6 months after the SA. The first one 7 days after the SA and the last one after 6 months. The first SMS (or mail or other new media) is sent soon after the SA because studies on adult suicide attempters underline the importance of an early start for the connectedness measures. The text messages are evolving in time, and are adapted to the genre of the adolescent.

The control arm is represented by the group CLASSIC with usual care.

Outcome measures Primary outcome The primary outcome is the delay of recurrence of suicide attempt during 6 months after the inclusion in the study. The recurrence and its date of occurrence will be collected by a member of the research team in each participating hospital.

Secondary outcomes The secondary outcomes include evaluation and evolution in a 6-month period after the SA of adolescent' social network using the Multidimensional Scale of Perceived Social Support (MSPSS), evaluation and evolution in a 6-month period after the SA of adolescent health-related quality of life using Kidscreen-27 and VSP-A, and evolution in a 6-month period after the SA of adolescent' depression using Center for Epidemiologic Studies Depression Scale (CES-D). The scores and their evolution will be compared between the groups CLASSIC and MEDIA.

The delay of recurrence of suicide attempt during 6 months after the end of the intervention by sending SMS (or mail or other new media). The recurrence and its date of occurrence will be collected by a member of the research team in each participating hospital.

The delay of death by suicide during 6 months after the end of the intervention. The suicide and its date of occurrence will be collected by a member of the research team in each participating hospital.

The number of callphone spent in the unit of care between adolescents of the group Media and those of the group Classic. They will be noted in a notebook planned for that purpose.

Instruments The text messages have been worked in focus group of peers and with adolescents. A pilot study has also been carried out in 2015 (MEDIADO) to refine their content. The text messages will be changing over time. They will be personalized with the surname of the patient and the name of the psychiatrist or his/her immediate superior who has met the patient after the SA. The number of the unit will be underlined in the message and the patient will be encouraged to call whenever he/she will feel the need to do it and will specify that someone will be always present for him/her.

The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item self-report with 5 possible answers by item. It assesses perceptions of social support from family members, friends, and significant others. It has been already used in other countries (29-30) and has been translated and validated in French by a team of Toulouse (31). The three subscales, each addressing a different source of support, were identified and found to have strong factorial validity. The MSPSS had also a good internal and test-retest reliability as well as moderate construct validity. High levels of perceived social support are associated with low levels of depression and anxiety.

The Kidscreen-27 is a 27-item self-report developed by an European group (32), validated in 12 European countries. It evaluates physical wellness, psychological wellness, relationships with parents, social network, relationships with friends, and schooling. The internal consistency is good as the discriminating power.

The VSP-A is a 37-item self-report with 10 dimensions, validated in French. This self-report has a good internal consistency as its construct validity and its content validity are also good (33).

The CES-D is a 12-item self report with a good internal consistency, validated in French.

The baseline personal, familial and social characteristics will be collected from medical records in order to explore factors that influence outcomes.

Statistical analyses The primary analyses will be conducted on an intention-to-treat basis using data for all randomized participants, although a per protocol analysis of the primary outcome will also be reported. There will be adjusted on the center. Continuous variables will be described with mean (and standard deviation) or median (and range), and categorical variables with number and percentage, as appropriate. The Chi-square or Fisher exact tests will be used for analysis of qualitative variables and the Student t or Mann-Whitney tests for quantitative variables.

Differences in both primary and secondary outcomes between the two groups of the study will be tested independently.

ELIGIBILITY:
Inclusion Criteria:

* be treated for a suicide attempt
* be 13-17 years old
* Patient living in the inter region or being able to be reorientated in the center of inclusion in case of recurrence of suicide attemps
* have consent of patient and his/her parents to participation in research.

Exclusion Criteria:

* The parents or/and patient who will refuse or who won't be able to accept to participate (somatic or understandability reasons),
* Incarcerated patient
* Those without any cell phone.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Delay of recurrence of suicide attempt | 6 months
  The primary outcome is the delay of recurrence of suicide attempt during 6 months after the inclusion in the study. The recurrence and its date of occurrence will be collected by a member of the research team in each participating hospital.

SECONDARY OUTCOMES:
Social Support | 6 months
  Evaluation and evolution in a 6-month period after the suicide attempt of adolescent' social network using the Multidimensional Scale of Perceived Social Support (MSPSS)
Quality of life | 6 months
  Evaluation and evolution in a 6-month period after the suicide attempt of adolescent health-related quality of life using Kidscreen-27 and VSP-A
Depression | 6 months
  Evaluation and evolution in a 6-month period after the suicide attempt of adolescent' depression using Center for Epidemiologic Studies Depression Scale (CES-D)
Delay of recurrence of suicide attempt | 6 to 12 months after suicide attempt
  Delay of recurrence of suicide attempt during 6 to 12 months after the inclusion in the study. The recurrence and its date of occurrence will be collected by a member of the research team in each participating hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne LIGIER, Dr, Study Director — Service de Psychiatrie de l'enfant et de l'adolescent, CHRU de Nancy; Catherine PICHENÉ, Dr, Principal Investigator — CPN, Unité d'Accueil des Urgences Psychiatriques; Philippe CHABERT, Dr, Principal Investigator — Unité de psychopathologie de l'adolescent Service Psychothérapique pour enfants et adolescents Pôle de Psychiatrie et Santé Mentale Hôpitaux Universitaires de Strasbourg; Sylvie NEZELOF, Dr, Principal Investigator — Service de Pédopsychiatrie Hôpital Jean Minjoz. CHRU de Besançon; Pascal PANNETIER, Dr, Principal Investigator — Service de Psychiatrie d'Urgence et de Liaison, dans les locaux du CHR Metz-Thionville Hôpital Mercy. CHR Metz-Thionville; Jean-Michel PINOIT, Dr, Principal Investigator — Service de Psychiatrie de l'enfant et de l'adolescent Hôpital d'enfants. CHU de Dijon; Anne-Catherine ROLLAND, Dr, Principal Investigator — Service de Psychothérapie de l'enfant et de l'adolescent Hôpital Robert Debré. CHU de Reims
Locations (5):
- France (5):
  - CHRU Besançon, Besançon
  - Hôpital de Mercy. CHR de Metz-Thionville, Metz
  - Chu Reims, Reims
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Centre Psychothérapique de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Study results will be restituted to each participant if they ask for it.

REFERENCES:
- [Background] 1. World Health Organization WHO. (2011). http://www.who.int/maternal_child_adolescent/topics/adolescence/fr/ Accessed April 2016
- [Background] Hawton K, Rodham K, Evans E, Weatherall R. Deliberate self harm in adolescents: self report survey in schools in England. BMJ. 2002 Nov 23;325(7374):1207-11. doi: 10.1136/bmj.325.7374.1207. PMID 12446536
- [Background] Moran P, Coffey C, Romaniuk H, Olsson C, Borschmann R, Carlin JB, Patton GC. The natural history of self-harm from adolescence to young adulthood: a population-based cohort study. Lancet. 2012 Jan 21;379(9812):236-43. doi: 10.1016/S0140-6736(11)61141-0. Epub 2011 Nov 16. PMID 22100201
- [Background] Wong JP, Stewart SM, Claassen C, Lee PW, Rao U, Lam TH. Repeat suicide attempts in Hong Kong community adolescents. Soc Sci Med. 2008 Jan;66(2):232-41. doi: 10.1016/j.socscimed.2007.08.031. Epub 2007 Oct 4. PMID 17919796
- [Background] Miranda R, Scott M, Hicks R, Wilcox HC, Harris Munfakh JL, Shaffer D. Suicide attempt characteristics, diagnoses, and future attempts: comparing multiple attempters to single attempters and ideators. J Am Acad Child Adolesc Psychiatry. 2008 Jan;47(1):32-40. doi: 10.1097/chi.0b013e31815a56cb. PMID 18174823
- [Background] Thompson MP, Light LS. Examining gender differences in risk factors for suicide attempts made 1 and 7 years later in a nationally representative sample. J Adolesc Health. 2011 Apr;48(4):391-7. doi: 10.1016/j.jadohealth.2010.07.018. Epub 2010 Oct 8. PMID 21402269
- [Background] MacDonald R, Taylor J, Clarke D. The relationship between early suicide behaviors and mental health: results from a nine-year panel study. J Adolesc. 2009 Oct;32(5):1159-72. doi: 10.1016/j.adolescence.2009.01.012. Epub 2009 Mar 9. PMID 19272640
- [Background] Ligier F, Guillemin F, Angot C, Bourion S, Kabuth B. Recurrence of suicide attempt in adolescents lost to contact early by clinicians: The 10-year REPEATERS cohort of French adolescents. J Adolesc. 2015 Aug;43:111-8. doi: 10.1016/j.adolescence.2015.05.011. Epub 2015 Jun 12. PMID 26073674
- [Background] Vaiva G, Jardon V, Vaillant A, Ducrocq F. [What can we do to prevent the suicide re-attempts?]. Rev Prat. 2011 Feb;61(2):202-3, 206-7. French. PMID 21618769
- [Background] Davidson K, Norrie J, Tyrer P, Gumley A, Tata P, Murray H, Palmer S. The effectiveness of cognitive behavior therapy for borderline personality disorder: results from the borderline personality disorder study of cognitive therapy (BOSCOT) trial. J Pers Disord. 2006 Oct;20(5):450-65. doi: 10.1521/pedi.2006.20.5.450. PMID 17032158
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] Weinberg I, Gunderson JG, Hennen J, Cutter CJ Jr. Manual assisted cognitive treatment for deliberate self-harm in borderline personality disorder patients. J Pers Disord. 2006 Oct;20(5):482-92. doi: 10.1521/pedi.2006.20.5.482. PMID 17032160
- [Background] Bateman A, Fonagy P. Effectiveness of partial hospitalization in the treatment of borderline personality disorder: a randomized controlled trial. Am J Psychiatry. 1999 Oct;156(10):1563-9. doi: 10.1176/ajp.156.10.1563. PMID 10518167
- [Background] Evans K, Tyrer P, Catalan J, Schmidt U, Davidson K, Dent J, Tata P, Thornton S, Barber J, Thompson S. Manual-assisted cognitive-behaviour therapy (MACT): a randomized controlled trial of a brief intervention with bibliotherapy in the treatment of recurrent deliberate self-harm. Psychol Med. 1999 Jan;29(1):19-25. doi: 10.1017/s003329179800765x. PMID 10077290
- [Background] Motto JA, Bostrom AG. A randomized controlled trial of postcrisis suicide prevention. Psychiatr Serv. 2001 Jun;52(6):828-33. doi: 10.1176/appi.ps.52.6.828. PMID 11376235
- [Background] 16. Beautrais AL, Gibb SJ, Faulkner A, Mulder RT. A randomised controlled trial of a brief intervention to reduce repeat presentations to the emergency department for suicide attempt. Annals of Emergency Medicine. 2008;51:474
- [Background] Carter GL, Clover K, Whyte IM, Dawson AH, D'Este C. Postcards from the EDge project: randomised controlled trial of an intervention using postcards to reduce repetition of hospital treated deliberate self poisoning. BMJ. 2005 Oct 8;331(7520):805. doi: 10.1136/bmj.38579.455266.E0. Epub 2005 Sep 23. PMID 16183654
- [Background] Vaiva G, Walter M, Al Arab AS, Courtet P, Bellivier F, Demarty AL, Duhem S, Ducrocq F, Goldstein P, Libersa C. ALGOS: the development of a randomized controlled trial testing a case management algorithm designed to reduce suicide risk among suicide attempters. BMC Psychiatry. 2011 Jan 2;11:1. doi: 10.1186/1471-244X-11-1. PMID 21194496
- [Background] Czyz EK, Liu Z, King CA. Social connectedness and one-year trajectories among suicidal adolescents following psychiatric hospitalization. J Clin Child Adolesc Psychol. 2012;41(2):214-26. doi: 10.1080/15374416.2012.651998. PMID 22417194
- [Background] Berrouiguet S, Alavi Z, Vaiva G, Courtet P, Baca-Garcia E, Vidailhet P, Gravey M, Guillodo E, Brandt S, Walter M. SIAM (Suicide intervention assisted by messages): the development of a post-acute crisis text messaging outreach for suicide prevention. BMC Psychiatry. 2014 Nov 18;14:294. doi: 10.1186/s12888-014-0294-8. PMID 25404215
- [Background] Milner AJ, Carter G, Pirkis J, Robinson J, Spittal MJ. Letters, green cards, telephone calls and postcards: systematic and meta-analytic review of brief contact interventions for reducing self-harm, suicide attempts and suicide. Br J Psychiatry. 2015 Mar;206(3):184-90. doi: 10.1192/bjp.bp.114.147819. PMID 25733570
- [Background] Brian RM, Ben-Zeev D. Mobile health (mHealth) for mental health in Asia: objectives, strategies, and limitations. Asian J Psychiatr. 2014 Aug;10:96-100. doi: 10.1016/j.ajp.2014.04.006. Epub 2014 Apr 27. PMID 25042960
- [Background] Collins JL, Champion JD. Assessment of mobile device and SMS Use for Diet and Exercise Information Among Rural Mexican-American adolescents. J Pediatr Nurs. 2014 Nov-Dec;29(6):493-502. doi: 10.1016/j.pedn.2014.03.020. Epub 2014 Mar 15. PMID 24704179
- [Background] 24. Gibson K, Cartwright C. Young people's experiences of mobile phone text counseling: Balancing connection and control. Child Youth Ser Rev. 2014;73:96-104
- [Background] Hawton K, Fagg J, Platt S, Hawkins M. Factors associated with suicide after parasuicide in young people. BMJ. 1993 Jun 19;306(6893):1641-4. doi: 10.1136/bmj.306.6893.1641. PMID 8324431
- [Background] Hinman RS, McCrory P, Pirotta M, Relf I, Crossley KM, Reddy P, Forbes A, Harris A, Metcalf BR, Kyriakides M, Novy K, Bennell KL. Efficacy of acupuncture for chronic knee pain: protocol for a randomised controlled trial using a Zelen design. BMC Complement Altern Med. 2012 Sep 19;12:161. doi: 10.1186/1472-6882-12-161. PMID 22992309
- [Background] Hatcher S, Sharon C, House A, Collins N, Collings S, Pillai A. The ACCESS study: Zelen randomised controlled trial of a package of care for people presenting to hospital after self-harm. Br J Psychiatry. 2015 Mar;206(3):229-36. doi: 10.1192/bjp.bp.113.135780. Epub 2015 Jan 22. PMID 25614531
- [Background] Adamson J, Cockayne S, Puffer S, Torgerson DJ. Review of randomised trials using the post-randomised consent (Zelen's) design. Contemp Clin Trials. 2006 Aug;27(4):305-19. doi: 10.1016/j.cct.2005.11.003. Epub 2006 Feb 7. PMID 16455306
- [Background] 29. Chou Kee-lee. Assessing Chinese adolescents' social support: the multidimensional scale of perceived social support. Pers Individ Dif. 2000;28: 299-307
- [Background] Osman A, Lamis DA, Freedenthal S, Gutierrez PM, McNaughton-Cassill M. The multidimensional scale of perceived social support: analyses of internal reliability, measurement invariance, and correlates across gender. J Pers Assess. 2014;96(1):103-12. doi: 10.1080/00223891.2013.838170. Epub 2013 Oct 3. PMID 24090236
- [Background] Denis A, Callahan S, Bouvard M. Evaluation of the French version of the multidimensional scale of perceived social support during the postpartum period. Matern Child Health J. 2015 Jun;19(6):1245-51. doi: 10.1007/s10995-014-1630-9. PMID 25366102
- [Background] 32. The KIDSCREEN Group Europe. The KIDSCREEN Questionnaires - Quality of life questionnaires for children and adolescents. Handbook. Lengerich: Pabst Science Publishers. 2006
- [Background] Sapin C, Simeoni MC, El Khammar M, Antoniotti S, Auquier P. Reliability and validity of the VSP-A, a health-related quality of life instrument for ill and healthy adolescents. J Adolesc Health. 2005 Apr;36(4):327-36. doi: 10.1016/j.jadohealth.2004.01.016. PMID 15780788
- [Background] Chabrol H, Montovany A, Chouicha K, Duconge E. [Study of the CES-D on a sample of 1,953 adolescent students]. Encephale. 2002 Sep-Oct;28(5 Pt 1):429-32. French. PMID 12386544
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Ligier F, Kabuth B, Guillemin F. MEDIACONNEX: a multicenter randomised trial based on short message service to reduce suicide attempt recurrence in adolescents. BMC Psychiatry. 2016 Jul 19;16:251. doi: 10.1186/s12888-016-0965-8. PMID 27435094